CLINICAL TRIAL: NCT04602793
Title: Sonographic Evaluation Of Nerve Thickness In Traumatic Lower-Limb Amputees: a Clinical and Sonographic-controlled Study
Brief Title: Sonographic Evaluation Of Nerve Thickness In Traumatic Lower-Limb Amputees
Status: Completed | Type: Observational
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Sefa Gümrük Aslan, Sonographic Evaluation Of Nerve Thickness In Traumatic Lower-Limb Amputees: a Clinical and Sonographic-controlled Study, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: 6
Record Dates: First submitted 2020-10-21; First posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Amputation, Traumatic
Keywords: Amputation; Prosthesis; peripheral nerves; ultrasonography
MeSH Terms: conditions — Amputation, Traumatic | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ultrasonography — All ultrasonographic examinations were performed by a single physiatrist experienced in musculoskeletal sonography. The full course of the sciatic nerve (SN), tibial nerve (TN), and common peroneal nerve (CPN) was assessed in a craniocaudal direction starting from the subgluteal fold to the popliteal fossa. The probe was placed axially on the nerves (perpendicular to the nerve) and the cross-sectional area (CSA) was measured at the same level proximal to the bifurcation for the SN , and at a point distal to the bifurcation of the SN for the TN and CPN (Figure 2). The values from the normal sides were accepted as controls.

SUMMARY:
Lower limb amputation (LLA) commonly affects young and active people who have long life expectancy. It is a major surgery causing many functional deficiencies which can reduce overall health quality and physical condition of the wounded persons and necessitating a multidisciplinary rehabilitation programme. High-frequency ultrasonography (US) is useful in evaluating peripheral nerves because of it has many superiority to other techniques. The advantages of US is; it has high resolution but no ionized radiation. It is possible to make dynamic and real-time imaging. It was showed that US have the same specificity and more sensitivity than magnetic resonance (MR) imaging in evaluating peripheral nerves. The aim of this study is to evaluate the sciatic, tibial and peroneal nerves of traumatic lower-limb amputees with the help of sonography and find the relationship between sonographic values and clinical characteristics.

DETAILED DESCRIPTION:
A total of thirty-three participants (age range 18-65) who had lower extremity amputation due to traumatic injury and were followed up in tertiary amputee clinic were included in this cross-sectional trial. The study was conducted between April 2019 and April 2020. Participants were totally volunteers and informed about the nature of the study. Written informed consent was obtained prior to assessment from all individuals. The study was conducted by the latest version of the principles of the Declaration of Helsinki protocol. All procedures were in consistency with the Helsinki Declarations of 1975. The study was approved by the local ethical committee.

All patients had completed stump healing. Patients with any disease affecting the peripheral nerves (eg, diabetes mellitus, infections, metabolic problems, inherited causes, and exposure to toxins) were excluded.

Demographic and clinical characteristics of the participants including age, gender, amputation findings (etiology, time since amputation, level, and side), prosthesis use findings (time since prosthesis use, daily use time, type, type of liner, prosthetic foot type), and functional K level of activity after amputation were recorded.

The presence, etiology, and duration of pain were questioned, and the intensity of pain was assessed by visual analog scale (VAS). Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) was used to evaluate neuropathic pain for the residual limb. The patient's satisfaction with the current prosthesis was evaluated numerically between 0 (not satisfied at all) and 10 (completely satisfied).

All ultrasonographic examinations were performed by a single physiatrist experienced in musculoskeletal sonography. A 5-12 MHz linear transducer (Logic e portable; GE Healthcare, China) was used. To optimize image quality, minimal pressure was applied to the transducer. Each examination was performed bilaterally while patients were in the prone position. The full course of the sciatic nerve (SN), tibial nerve (TN), and common peroneal nerve (CPN) was assessed in a craniocaudal direction starting from the subgluteal fold to the popliteal fossa. The probe was placed axially on the nerves (perpendicular to the nerve) and the cross-sectional area (CSA) was measured at the same level proximal to the bifurcation for the SN (Figure 1), and at a point distal to the bifurcation of the SN for the TN and CPN (Figure 2). The values from the normal sides were accepted as controls. The presence of a neuroma was also evaluated throughout the nerve, particularly at the distal ends.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-65
* Patients who have been followed up for at least 3 months with the diagnosis of unilateral transtibial amputation
* Patients who have been using prostheses for at least 3 months

Exclusion Criteria:

* Bilateral amputation
* Previous history of any trauma/surgical history of the lower extremities (other than amputation)
* Rheumatic diseases
* Contracture of the knee and the ankle of the intact limb .Presence of comorbid diseases that may cause peripheral nerve lesions ( e.g diabetis mellitus, using alcohol, thyroid diseases...)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of thirty-three participants (age range 18-65) who had lower extremity amputation due to traumatic injury and were followed up in tertiary amputee clinic were included in this cross-sectional trial. All patients had completed stump healing. Patients with any disease affecting the peripheral nerves (eg, diabetes mellitus, infections, metabolic problems, inherited causes, and exposure to toxins) were excluded.
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Sciatic nerve (SN), tibial nerve (TN), and common peroneal nerve (CPN) thickness measurements | through study completion, an average of one and a half months]
  Sciatic nerve (SN), tibial nerve (TN), and common peroneal nerve (CPN) thickness and cross sectional area measurements will be performed by using ultrasound.

SECONDARY OUTCOMES:
Visual analog scale (VAS) | through study completion, an average of one and a half months
  The Visual analog scale (VAS) will be used for the assessment of the intensity of pain
Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) | through study completion, an average of one and a half months
  The Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) will be used to evaluate neuropathic pain for the residual limb.

CONTACTS AND LOCATIONS:
Overall Officials: sefa Gümrük Aslan, MD, Principal Investigator — Gaziler PMR, Training and Research Hospital, Department of PMR
Locations (1):
- Gaziler PMR, Training and Research Hospital, Department of PMR, Ankara, Çankaya/turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No